CLINICAL TRIAL: NCT02868892
Title: A Phase II Study of Pemetrexed in Recurrent Cervical Adenocarcinomas
Brief Title: A Study of Pemetrexed in Recurrent Cervical Adenocarcinomas
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: departure of PI from institution and poor population for study participation
Sponsor: Western Regional Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CWG2014034 Pemetrexed Cervica
Record Dates: First submitted 2016-05-02; First posted 2016-08-16 (Estimated); Results first posted 2018-11-02 (Actual); Last update posted 2018-11-02 (Actual); Status verified 2018-10

CONDITIONS: Adenocarcinoma of the Cervix; Adenosquamous Cell Carcinoma of the Cervix
MeSH Terms: interventions — Pemetrexed

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Pemetrexed (Experimental): Pemetrexed 500 mg/m2 will be administered on an outpatient basis on an every three week schedule. Pemetrexed will be administered as a 10 minutes intravenous (IV) infusion in (for 500-mg vial) 100 ml of saline via peripheral vein or central line on Day 1 of each 21 day cycle.
  Interventions: Drug: Pemetrexed

INTERVENTIONS:
Drug: Pemetrexed — Pemetrexed 500 mg/m2
  Other Names: Alimta

SUMMARY:
Patients with advanced or recurrent adenocarcinoma or adenosquamous cell carcinoma of the cervix will receive Pemetrexed.

DETAILED DESCRIPTION:
Patients will receive Pemetrexed 500 mg/m2 every three week.

On initiation of pemetrexed, on day one of first chemotherapy cycle, patients will begin taking folic acid at a dose of 350 to 600 mcg daily as well as receive an intramuscular injection of 1000 mcg of vitamin B12, with subsequent vitamin B12 injections given every 9 weeks while on study.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have had advanced or recurrent adenocarcinoma or adenosquamous cell carcinoma of the cervix with documented disease progression
2. Patients must have had measurable disease defined as at least one lesion that could be accurately measured in at least one dimension, which must have been 20 mm when measured by conventional techniques including palpation, plain X-ray, computerized tomography (CT), and magnetic resonance imaging(MRI) or 10 mm when measured by spiral CT
3. 18 years of age or older
4. Eastern Cooperative Oncology Group (ECOG) performance status score < 2 and a life expectancy >3 months
5. Life expectancy ≥ 12 weeks
6. Participants must have measureable disease by RECIST criteria
7. Absolute neutrophil count > 1500 mm3, platelet count ≥ 100×109 L, hemoglobin ≥ 8.5 g/dL
8. Creatinine clearance ≥ 45 mL/min using the standard Cockcroft and Gault formula (below) or glomerular filtration rate (GFR) measured by Tc99m-diethylenetriaminepentacetate (DPTA) serum clearance method:

   1. Males: [140 - Age in years] × Actual Body Weight (kg) 72 × Serum Creatinine (mg/dL)
   2. Females: Estimated creatinine clearance for males × 0.85
9. Total bilirubin ≤ 2 mg/dL, aspartate transaminase (AST) and alanine transaminase (ALT) AST/ALT ≤ 5 times the upper limit of normal range
10. At least 21 days from administration of chemotherapy
11. No remaining grade 2 or higher toxicity from prior cancer therapies unless judged to be clinically insignificant by the Principal Investigator
12. At least four (4) weeks from prior major surgery
13. Willingness to provide permission to access archived tumor samples and additional blood samples for evaluation of Foundation One Analysis where available Enterprise wide.
14. Women of child-bearing potential (i.e., women who are pre-menopausal or not surgically sterile) must be willing to use an acceptable contraceptive method (abstinence, oral contraceptive or double barrier method) for the duration of the study and for 30 days following the last dose of study drug, and must have a negative urine or serum pregnancy test within 2 weeks prior to beginning treatment on this trial.

Exclusion Criteria:

1. Uncontrolled cardiac disease, congestive heart failure, angina, arrhythmias or hypertension.
2. Myocardial infarction or unstable angina within 2 months of treatment.
3. Known human immunodeficiency virus (HIV) infection or chronic active Hepatitis B or C (patients are NOT required to be tested for the presence of such viruses prior to therapy on this protocol).
4. Active clinically serious infection > CTCAE (version 4.03) Grade 2.
5. Thrombotic or embolic events such as a cerebrovascular accident including transient ischemic attacks within the past 6 months.
6. Pulmonary hemorrhage/bleeding event ≥ CTCAE Grade 2 within 4 weeks of first dose of study drug.
7. Any other hemorrhage/bleeding event ≥ CTCAE Grade 3 within 4 weeks of first dose of study drug.
8. Serious non-healing wound, ulcer, or bone fracture.
9. Major surgery, open biopsy or significant traumatic injury within 4 weeks of first study drug.
10. Inability to complete informed consent process and adhere to the protocol treatment plan and follow-up requirements.
11. Concurrent severe illness such as active infection, or psychiatric illness/social situations that would limit safety and compliance with study requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2015-07; Primary Completion 2017-07 (Actual); Study Completion 2017-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Farley, MD, Principal Investigator — Western Regional Medical Center
Locations (1):
- Western Regional Medical Center, Inc., Goodyear, Arizona, United States

IPD SHARING:
Plan to Share IPD: Yes
Plan to present data as abstract format

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Pemetrexed
Started | 6
Completed | 0
Not Completed | 6
Not completed — Investigator left site and no follow-up | 6

BASELINE CHARACTERISTICS:
Arm/Group | Pemetrexed
Number analyzed (Participants) | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 6
  >=65 years | 0
Age, Continuous [Mean (Full Range); unit: years] | 54 [37 to 58]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 1
  Unknown or Not Reported | 3
Region of Enrollment [Number; unit: participants]
  United States | 6

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival
Description: Evaluate the progression free survival of recurrent cervical adenocarcinoma. Progression-Free Survival is defined as the period of time from the date of first study drug administration to the date that the subject is determined to have progressive disease or death due to any cause.
Time Frame: 2 years
Population: Investigator no longer at site. Study was closed with no PI transfer, data collection or statistical analysis.
Arm/Group | Pemetrexed
Number analyzed (Participants) | 0

2. Secondary Outcome: Response Rate
Description: Evaluate the response rate for recurrent cervical adenocarcinomas treated with pemetrexed. Measurable disease is defined as at least one lesion that can be accurately measured in at least one dimension which must have been 20 mm when measured by conventional techniques including palpation, plain X-ray, CT, and MRI or 10 mm when measured by spiral CT.
Time Frame: 2 years
Population: Investigator no longer at site. Study was closed with no PI transfer, data collection or statistical analysis.
Arm/Group | Pemetrexed
Number analyzed (Participants) | 0

3. Secondary Outcome: Overall Survival
Description: Evaluate Overall survival for recurrent cervical adenocarcinomas treated with pemetrexed.
Time Frame: 2 years
Population: Investigator no longer at site. Study was closed with no PI transfer, data collection or statistical analysis.
Arm/Group | Pemetrexed
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 6-12 months
Arm/Group | Pemetrexed
All-Cause Mortality (participants affected / at risk) | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6
Other Adverse Events (participants affected / at risk) | 0/6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-03-29): https://cdn.clinicaltrials.gov/large-docs/92/NCT02868892/Prot_SAP_000.pdf